CLINICAL TRIAL: NCT04800107
Title: Effect of Highly Bioavailable Curcumin on Subjective Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1682516
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Tinnitus, Subjective
Keywords: Curcumin; Anti-inflammatory compound; Turmeric
MeSH Terms: conditions — Tinnitus | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized to a treatment or placebo group after completing both the TFI and THI surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Subjects will be provided with a supply of capsules containing 500 mg of curcumin-phosphatidylcholine combined with 250 mg of boswellia-phosphatidyl. Subjects will take 1 capsule by mouth twice daily for 30 days.
  Interventions: Biological: Curcumin-phosphatidylcholine
- Placebo Group (Placebo Comparator): Subjects will be provided with a placebo compound with instructions to take 1 capsule by mouth twice daily for 30 days.
  Interventions: Biological: Placebo capsule

INTERVENTIONS:
Biological: Curcumin-phosphatidylcholine — 500 mg of curcumin-phosphatidylcholine combined with 250 mg of boswellia-phosphatidyl
  Other Names: Tumeric
  Arms: Treatment Group
Biological: Placebo capsule — Placebo capsule
  Arms: Placebo Group

SUMMARY:
This study will assess the effectiveness of highly bioavailable curcumin in suppressing subjective tinnitus based on pre- and post-treatment evaluations using the validated Tinnitus Functional Index (TFI) and Tinnitus Handicap Inventory (THI) surveys.

DETAILED DESCRIPTION:
Subjects with severe, subjective tinnitus due to sensorineural hearing loss will complete both TFI and THI surveys prior to starting therapy. Subjects will then be randomized to a treatment or placebo group. The treatment group will be provided with a supply of capsules containing 500 mg of curcumin-phosphatidylcholine combined with 250 mg of boswellia-phosphatidylcholine, which increases curcumin bioavailability. Subjects in the treatment arm will be instructed to take 1 capsule by mouth twice daily for 30 days. Placebo group subjects will be provided with a placebo compound with instructions to take the same number of capsules by mouth for the same period of time. Both the active compound and the placebo will be provided by Smartceuticals, Inc (910 W. Van Buren St. Ste 100-376 Chicago, IL 60607) to the outpatient pharmacy at Ascension Providence Park (Novi, MI), which will be responsible for storage, distribution and tracking. After 30 days, patients will be asked to return bottles to the pharmacy with any unused capsules to confirm and monitor compliance. Placebo and active agent capsules and bottles will be identical in appearance with the exception of a unique alphanumeric code on the bottle label that identifies whether the distributed capsules contain active agent or placebo. This code will be matched to the participating subject by the pharmacy and will be used at the end of the study to determine which treatment arm each subject was in. To facilitate blinding, the master list of alphanumeric codes will be maintained by the manufacturer. At the completion of therapy, subjects from both groups will re-take the TFI and THI.

ELIGIBILITY:
Inclusion Criteria:

* Adults with subjective tinnitus due to sensorineural hearing loss as determined by routine audiogram.

Exclusion Criteria:

* Adults with subjective tinnitus due to another cause
* Sensitivity or allergy to test compounds
* Use of other off-label medications, substances, treatments specifically for tinnitus mitigation (e.g., anti-depressant/anxiety medications, GABA-inhibitors, psychiatric-based interventions/counseling)
* Pregnancy
* Patients taking anticoagulants to minimize risk of drug-drug interactions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change on the Tinnitus Functional Index (TFI) | Evaluate at the beginning of the trial and at the end of the 30 day treatment period.
  Administer the TFI survey

SECONDARY OUTCOMES:
Determine Changes in the Tinnitus Handicap Inventory (THI) | Evaluate at the beginning of the trial and at the end of the 30 day treatment period.
  Measure the Tinnitus Handicap Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Seilish Babu, MD, Principal Investigator — Michigan Ear Institute
Locations (3):
- United States (3):
  - Michigan Ear Institute, Farmington Hills, Michigan
  - Michigan Ear Institute, Novi, Michigan
  - Michigan Ear Institute, Royal Oak, Michigan

REFERENCES:
- [Background] Soyalic H, Gevrek F, Karaman S. Curcumin protects against acoustic trauma in the rat cochlea. Int J Pediatr Otorhinolaryngol. 2017 Aug;99:100-106. doi: 10.1016/j.ijporl.2017.05.029. Epub 2017 Jun 5. PMID 28688549
- [Background] Haryuna TS, Riawan W, Nasution A, Ma'at S, Harahap J, Adriztina I. Curcumin Reduces the Noise-Exposed Cochlear Fibroblasts Apoptosis. Int Arch Otorhinolaryngol. 2016 Oct;20(4):370-376. doi: 10.1055/s-0036-1579742. Epub 2016 Mar 4. PMID 27746842
- [Background] Soyalic H, Gevrek F, Koc S, Avcu M, Metin M, Aladag I. Intraperitoneal curcumin and vitamin E combination for the treatment of cisplatin-induced ototoxicity in rats. Int J Pediatr Otorhinolaryngol. 2016 Oct;89:173-8. doi: 10.1016/j.ijporl.2016.08.012. Epub 2016 Aug 24. PMID 27619052
- [Background] Mirzaei H, Shakeri A, Rashidi B, Jalili A, Banikazemi Z, Sahebkar A. Phytosomal curcumin: A review of pharmacokinetic, experimental and clinical studies. Biomed Pharmacother. 2017 Jan;85:102-112. doi: 10.1016/j.biopha.2016.11.098. Epub 2016 Dec 5. PMID 27930973
- [Background] Yamaguchi T, Yoneyama M, Onaka Y, Imaizumi A, Ogita K. Preventive effect of curcumin and its highly bioavailable preparation on hearing loss induced by single or repeated exposure to noise: A comparative and mechanistic study. J Pharmacol Sci. 2017 Aug;134(4):225-233. doi: 10.1016/j.jphs.2017.07.003. Epub 2017 Aug 8. PMID 28826625
- [Background] Gupta SC, Patchva S, Aggarwal BB. Therapeutic roles of curcumin: lessons learned from clinical trials. AAPS J. 2013 Jan;15(1):195-218. doi: 10.1208/s12248-012-9432-8. Epub 2012 Nov 10. PMID 23143785
- [Background] Castaneda R, Natarajan S, Jeong SY, Hong BN, Kang TH. Traditional oriental medicine for sensorineural hearing loss: Can ethnopharmacology contribute to potential drug discovery? J Ethnopharmacol. 2019 Mar 1;231:409-428. doi: 10.1016/j.jep.2018.11.016. Epub 2018 Nov 12. PMID 30439402
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Zeman F, Koller M, Figueiredo R, Aazevedo A, Rates M, Coelho C, Kleinjung T, de Ridder D, Langguth B, Landgrebe M. Tinnitus handicap inventory for evaluating treatment effects: which changes are clinically relevant? Otolaryngol Head Neck Surg. 2011 Aug;145(2):282-7. doi: 10.1177/0194599811403882. PMID 21493265